CLINICAL TRIAL: NCT01336894
Title: A Randomized Phase III Study of Sublobar Resection (+/- Brachytherapy) Versus Stereotactic Body Radiation Therapy in High Risk Patients With Stage I Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Surgery With or Without Internal Radiation Therapy Compared With Stereotactic Body Radiation Therapy in Treating Patients With High-Risk Stage I Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: recruiting or enrolling participants has halted prematurely and will not resume; participants are no longer being examined or treated
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z4099; U10CA076001 (NIH); NCI-2011-02667 (Registry Identifier: NCI Clinical Trials Reporting Office); CDR0000698986 (Registry Identifier: Physician Data Query)
Record Dates: First submitted 2011-04-15; First posted 2011-04-18 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Lung Cancer
Keywords: stage IA non-small cell lung cancer; stage IB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Iodine-125; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (SR+Brachytherapy) (Active Comparator): Patients undergo sublobar resection comprising either a wedge resection or anatomical segmentectomy with or without intraoperative brachytherapy comprising an iodine I 125 implant at the resection margin.
  Interventions: Procedure: therapeutic conventional surgery; Radiation: iodine I 125
- Arm II (SBRT) (Experimental): Patients undergo 3 fractions of stereotactic body radiation therapy at 2-8 days apart.
  Interventions: Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Undergo surgery
  Arms: Arm I (SR+Brachytherapy)
Radiation: iodine I 125 — Undergo seed implant radiotherapy
  Arms: Arm I (SR+Brachytherapy)
Radiation: stereotactic body radiation therapy — Undergo radiotherapy
  Arms: Arm II (SBRT)

SUMMARY:
RATIONALE: Surgery with or without internal radiation therapy may be an effective treatment for non-small cell lung cancer. Internal radiation uses radioactive material placed directly into or near a tumor to kill tumor cells. Stereotactic body radiation therapy may be able to send x-rays directly to the tumor and cause less damage to normal tissue. It is not yet known whether stereotactic body radiation therapy is more effective than surgery with or without internal radiation therapy in treating non-small cell lung cancer.

PURPOSE: This randomized phase III trial is studying how well surgery with or without internal radiation therapy works compared with stereotactic body radiation therapy in treating patients with high-risk stage IA or stage IB non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To ascertain whether patients treated by stereotactic body radiation therapy (SBRT) have a 3-year overall survival (OS) rate that is no more than 10% less than patients treated with sublobar resection (SR).

Secondary

* To compare loco-regional recurrence-free survival between study arms.
* To compare disease-free survival between study arms.
* To compare grade 3 or higher specific adverse event profiles between study arms at 1, 3, 6, and 12 months post-therapy.
* To compare pulmonary function between patients treated with SBRT and patients treated with SR.
* To compare the adverse events and pulmonary function tests (PFTs) in each arm for patients with low or high Charlson comorbidity index scores, including a test interaction between Charlson comorbidity index scores (low vs high) and treatment arm.

Tertiary

* To compare the quality-adjusted survival between the SBRT and SR treatments in terms of time to death (primary) and time until recurrence (secondary).
* To examine whether pre-operative and post-operative clinically significant deficits in previously identified prognostic PRO domains (overall quality of life [QOL], fatigue, anxiety, and dyspnea) are associated with shorter patient survival in this patient population and to compare the relative effectiveness of each treatment (SBRT and SR).
* To contribute to an ACOSOG bank of normative data in order to improve short/long-term outcomes of cancer patients by identifying patients experiencing clinically significant deficits in patient-reported outcomes and the relationship to genetic variables.
* To explore whether blood-based biomarkers, including osteopontins, will be able to predict which patients will be at high risk for recurrence by treatment with either SBRT or SR. (exploratory)
* To explore whether blood-based biomarkers, including TGF-β1, will be able to predict which patients will be at high risk for pulmonary complications by treatment with either SBRT or SR. (exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to planned brachytherapy (yes vs no) and ECOG performance status (0 vs 1 vs 2). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo sublobar resection comprising either a wedge resection or anatomical segmentectomy with or without intraoperative brachytherapy* comprising an iodine I 125 implant at the resection margin.
* Arm II: Patients undergo 3 fractions of stereotactic body radiation therapy at 2-8 days apart.

NOTE: *Patients may receive brachytherapy at the discretion of treating physician.

Patients may undergo blood sample collection at baseline and periodically during study for correlative studies. Tumor tissue samples may also be collected from patients who undergo resection.

Patients complete the Lung Cancer Symptom Scale (LCSS), the Linear Analogue Self-Assessment (LASA), and the UCDS Shortness of Breath quality-of-life questionnaires at baseline and periodically during study and follow-up.

After completion of study treatment, patients are followed up for 30 days, every 3 months for 2 years, every 6 months for 1 year, and then yearly for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Lung nodule suspicious for non-small cell lung cancer (NSCLC)

  * Biopsy confirmation is strongly recommended but not required; if biopsy is attempted and non-diagnostic, if the patient refuses biopsy, or if the risk of biopsy is considered too high, patients may be enrolled if the mass is suspicious for NSCLC based on two or more of the following criteria:

    * Positive smoking history
    * Absence of benign calcifications within suspicious nodule
    * Activity on PET greater than normal tissue
    * Evidence of growth compared to previous imaging
    * Presence of spiculation
* Tumor ≤ 4 cm maximum diameter, clinical stage IA or selected IB (i.e., with visceral pleural involvement) by PET/CT scan of the chest and upper abdomen performed within 60 days prior to registration
* All clinically suspicious mediastinal N1, N2, or N3 lymph nodes (> 1 cm short-axis dimension on CT scan and/or positive on PET scan) confirmed negative for involvement with NSCLC by one of the following methods: mediastinoscopy, anterior mediastinotomy, endoscopic and/or endobronchial ultrasonography (EUS/EBUS)-guided needle aspiration, CT-guided, or video-assisted thoracoscopic or open lymph node biopsy
* Tumor verified by a thoracic surgeon to be in a location that will permit sublobar resection
* Tumor located peripherally within the lung, defined as not touching any surface within 2 cm of the proximal bronchial tree in all directions

  * Patients with non-peripheral (central) tumors are NOT eligible
* No evidence of distant metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0, 1, or 2
* Patient at high-risk for surgery by meeting a minimum of one major criteria or two minor criteria as described below:

  * Major criteria

    * FEV1 ≤ 50% predicted
    * DLCO ≤ 50% predicted
  * Minor criteria

    * Age ≥ 75 years
    * FEV1 51-60% predicted
    * DLCO 51-60% predicted
    * Pulmonary hypertension (defined as a pulmonary artery systolic pressure greater than 40 mm Hg) as estimated by echocardiography or right heart catheterization
    * Poor left ventricular function (defined as an ejection fraction of 40% or less)
    * Resting or exercise arterial pO2 ≤ 55 mm Hg or SpO2 ≤ 88%
    * pCO2 > 45 mm Hg
    * Modified Medical Research Council (MMRC) Dyspnea Scale ≥ 3
* Not pregnant or nursing
* Negative urine or serum pregnancy test
* Fertile patients must use effective contraception
* No prior invasive malignancy, unless disease-free for ≥ 3 years prior to registration (except non-melanoma skin cancer, in-situ cancers).

PRIOR CONCURRENT THERAPY:

* No prior intra-thoracic radiotherapy

  * Prior radiotherapy as part of treatment for head and neck, breast, or other non-thoracic cancer is permitted
* Prior chemotherapy or surgical resection for the lung cancer being treated on this protocol is NOT permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2017-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiran C. Fernando, MD, Principal Investigator — Boston Medical Center
Locations (53):
- United States (49):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - University of California Davis Cancer Center, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Tufts Medical Center Cancer Center, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Baylor University Medical Center - Dallas, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
- Canada (4):
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec

REFERENCES:
- [Result] Fernando HC, Timmerman R. American College of Surgeons Oncology Group Z4099/Radiation Therapy Oncology Group 1021: a randomized study of sublobar resection compared with stereotactic body radiotherapy for high-risk stage I non-small cell lung cancer. J Thorac Cardiovasc Surg. 2012 Sep;144(3):S35-8. doi: 10.1016/j.jtcvs.2012.06.003. Epub 2012 Jul 11. PMID 22795435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirteen (13) participants were accrued between August 2011 and January 2013. The study was terminated prematurely on May 15, 2013 due to lack of accrual. No further follow up data are expected as of that date.
Pre-assignment Details: Two participants on Arm I refused/withdrew prior to beginning of protocol interventions. These two participants were excluded from all analyses.
Groups:
- Arm I (SR+Brachytherapy): Patients undergo sublobar resection (SR) comprising either a wedge resection or anatomical segmentectomy with or without intraoperative brachytherapy comprising an iodine I 125 implant at the resection margin.
- Arm II (SBRT): Patients undergo 3 fractions of stereotactic body radiation therapy (SBRT) at 2-8 days apart.
Period: Protocol Interventions
Arm/Group | Arm I (SR+Brachytherapy) | Arm II (SBRT)
Started | 4 | 7
Completed | 4 | 7
Not Completed | 0 | 0
Period: Follow-up
Arm/Group | Arm I (SR+Brachytherapy) | Arm II (SBRT)
Started | 4 | 7
Completed | 2 | 0
Not Completed | 2 | 7
Not completed — Study terminated prematurely | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (SR+Brachytherapy) | Arm II (SBRT) | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Median (Full Range); unit: years] | 65 [50 to 72] | 68 [53 to 81] | 68 [50 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 7 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 2 | 2
  United States | 4 | 5 | 9
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants]
  0=Asymptomatic and fully active | 2 | 3 | 5
  1=Symptomatic and fully ambulatory | 2 | 4 | 6
Institutional intent to use brachytherapy [Count of Participants; unit: Participants]
  Yes | 1 | 2 | 3
  No | 3 | 5 | 8
Baseline diffusing capacity of the lung for carbon monoxide (DLCO) [Median (Full Range); unit: Percentage of predicted] | 46 [33 to 80] | 43 [28 to 92] | 44 [28 to 92]
Baseline Forced Expiratory Volume in 1 second (FEV1) [Median (Full Range); unit: Percentage of predicted] | 42 [22 to 65] | 92 [44 to 118] | 54 [22 to 118]

OUTCOME MEASURES:

1. Primary Outcome: 3-year Overall Survival (OS) Rate
Description: Overall survival is defined as the time from randomization until death from any cause.
Time Frame: Up to 3 years post-randomization
Population: Study terminated prematurely. Planned analyses was not performed due to the nature of the closure endpoint data is not available.
Arm/Group | Arm I (SR+Brachytherapy) | Arm II (SBRT)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Loco-regional Recurrence-free Survival
Description: Loco-regional recurrence is defined as recurrence within the same lobe or hilum (N1 nodes), or within 2 cm of the staple line or within 2 cm of the PTV after treatment effects such as scarring have subsided.
Time Frame: Up to 5 years post-randomization
Population: as for outcome 1
Arm/Group | Arm I (SR+Brachytherapy) | Arm II (SBRT)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Adverse Event Profiles at 1 Month Post-therapy
Description: Adverse events are described and graded using the terminology and grading categories defined in the NCI's Common Toxicity Criteria (CTCAE), Version 4.0.
  Grading: Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening, Grade 5=Death.
Time Frame: 1 month post-therapy
Population: All enrolled participants who received protocol interventions and had adverse events reported at 1 month post-therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (SR+Brachytherapy) | Arm II (SBRT)
Number analyzed (Participants) | 4 | 7
Participants
  Chest wall pain: Grade 0 | 3 | 7
  Chest wall pain: Grade 1 | 1 | 0
  Chest wall pain: Grade 2 | 0 | 0
  Cough: Grade 0 | 3 | 5
  Cough: Grade 1 | 1 | 2
  Cough: Grade 2 | 0 | 0
  Dyspnea: Grade 0 | 4 | 6
  Dyspnea: Grade 1 | 0 | 1
  Dyspnea: Grade 2 | 0 | 0
  Hoarness: Grade 0 | 4 | 6
  Hoarness: Grade 1 | 0 | 1
  Hoarness: Grade 2 | 0 | 0
  Hypoxia: Grade 0 | 3 | 7
  Hypoxia: Grade 1 | 0 | 0
  Hypoxia: Grade 2 | 1 | 0
  Fatigue: Grade 0 | 4 | 6
  Fatigue: Grade 1 | 0 | 0
  Fatigue: Grade 2 | 0 | 1

4. Secondary Outcome: Adverse Event Profiles at 3 Months Post-therapy
Description: as for outcome 3
Time Frame: 3 months post-therapy
Population: All enrolled participants who received protocol interventions and had adverse event reported at months 3 post-therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (SR+Brachytherapy) | Arm II (SBRT)
Number analyzed (Participants) | 4 | 6
Participants
  Cough: Grade 0 | 3 | 4
  Cough: Grade 1 | 1 | 2
  Cough: Grade 2 | 0 | 0
  Hypoxia: Grade 0 | 3 | 6
  Hypoxia: Grade 1 | 0 | 0
  Hypoxia: Grade 2 | 1 | 0

5. Secondary Outcome: Adverse Event Profiles at 12 Months Post-therapy
Description: as for outcome 3
Time Frame: 12 months post-therapy
Population: as for outcome 1
Arm/Group | Arm I (SR+Brachytherapy) | Arm II (SBRT)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Disease-free Survival
Description: Disease free survival is defined as the time from randomization until documented disease recurrence or death, whichever occurs first. Patient who are disease free and alive at the time of analysis will be censored at the time of their last follow up.
Time Frame: Up to 5 years post-randomization
Population: as for outcome 1
Arm/Group | Arm I (SR+Brachytherapy) | Arm II (SBRT)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pulmonary Function Test Values
Description: Pulmonary function test values include forced expiratory volume 1 (FEV1), carbon monoxide diffusion (DLCO) and forced vital capacity (FVC).
Time Frame: Up to 12 months post-therapy
Population: as for outcome 1
Arm/Group | Arm I (SR+Brachytherapy) | Arm II (SBRT)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events reported since the participants received the study interventions to the date the study was closed prematurely on May 15, 2013 with no further follow up expected; up to 2 years from the start of the study.
Description: Adverse events are described and graded using the terminology and grading categories defined in the NCI's Common Toxicity Criteria (CTCAE), Version 4.0. Please note that the death NOS reported fell outside of the reporting window and was queried on but since the trial was terminated midstream the data management was not completed.
Arm/Group | Arm I (SR+Brachytherapy) | Arm II (SBRT)
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/7
Other Adverse Events (participants affected / at risk) | 3/4 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (SR+Brachytherapy) (N=4) | Arm II (SBRT) (N=7)
Death NOS (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (SR+Brachytherapy) (N=4) | Arm II (SBRT) (N=7)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (2) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Carbon monoxide diffusing capacity decreased (Investigations) | 0 (0) | 1 (1)
Forced expiratory volume decreased (Investigations) | 0 (0) | 1 (1)
Vital capacity abnormal (Investigations) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (8) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less